CLINICAL TRIAL: NCT00527254
Title: Telemedicine Influence in the Follow up of the Type 2 Diabetes Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Province of Malaga Health Department (Other Government)
Collaborators: Roche Diabetes Care (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TeleDiabecom 200501
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Type 2 Diabetes; Telemedicine; Self Monitoring Blood Glucose; Primary Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention)
- Telemedicine group (Active Comparator)
  Interventions: Device: Telemedicine system

INTERVENTIONS:
Device: Telemedicine system — Possibility of sending the SMBG values of the patients to a web page via phone mobile sms messages. The HCP had a password access to this web page to check the blood glucose values of the patients and if necessary send to them sms messages with recommendations.
  Arms: Telemedicine group

SUMMARY:
The purpose of this study is to evaluate the impact of a a real time teleassistance system in the clinical evolution of type 2 diabetic patients on self monitoring blood glucose in the Public National Primary Care System.

DETAILED DESCRIPTION:
The UKPDS study in type 2 diabetes and the DCCT in type 1, showed that intensive blood glucose control and the following HBA1c decrease were associated with a decrease of diabetic complications. Introducing telecontrol elements in the real time follow up of the patients, should help to know continuously patient blood glucose profile and add if necessary immediately therapeutical variations, to maintain HbA1c levels as low as possible.

The study compares type 2 diabetes patients performing self monitoring of blood glucose, followed up by their family doctor in their primary care unit with the extra support of a real time teleassistance system with type 2 diabetes patients performing self monitoring of blood glucose, followed up by their family doctor in their primary care unit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 Diabetes
* on SMBG al least 6 months before
* age superior of 30 years
* controlled in province of Málaga Primary Care Units

Exclusion Criteria:

* having diabetic complications or other diseases that could make difficult to use the telemedicine system
* patients who need a carer
* not passing the initial training (low cultural level)
* living in an area without mobile phone coverage

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2003-10; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
HBA1c Glycosylated hemoglobin | one year for every patient

SECONDARY OUTCOMES:
Blood glucose, Total Cholesterol, HDL Cholesterol,LDL Cholesterol, Triglycerides, BMI, systolic and diastolic blood pressure and system adherence | one year for every patient

CONTACTS AND LOCATIONS:
Overall Officials: Maria Isabel Rodríguez Idígoras, Doctor, Principal Investigator — Málaga Health Department (Junta de Andalucia)
Locations (1):
- Province of Malaga Health Department, Málaga, Málaga, Spain

REFERENCES:
- [Derived] Rodriguez-Idigoras MI, Sepulveda-Munoz J, Sanchez-Garrido-Escudero R, Martinez-Gonzalez JL, Escolar-Castello JL, Paniagua-Gomez IM, Bernal-Lopez R, Fuentes-Simon MV, Garofano-Serrano D. Telemedicine influence on the follow-up of type 2 diabetes patients. Diabetes Technol Ther. 2009 Jul;11(7):431-7. doi: 10.1089/dia.2008.0114. PMID 19580356